CLINICAL TRIAL: NCT05308732
Title: Phase I Study of Multiple Ascending Dose, to Investigate the Safety and Tolerability of the Use of Copaiba in Patients With Oral Cancer Submitted to Radiotherapy
Brief Title: Safety and Tolerability of the Use of Copaiba in Patients With Oral Cancer Submitted to Radiotherapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 34635020.5.0000.5274
Record Dates: First submitted 2020-08-06; First posted 2022-04-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Neoplasms; Mucositis Oral; Radiotherapy; Complications
Keywords: Head and Neck Neoplasms; Mucositis Oral; Radiotherapy; Complications
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis

STUDY DESIGN:
Intervention Model Description: The investigator will assign a unique number to the patient being evaluated to participate in the study. The patients included in the study will receive instructions on oral hygiene and the aqueous copaiba solution for mouthwash.
  The recruitment and design of the study will be carried out according to the "3 + 3" design (modified Fibonacci design) with the planned inclusion of 6 successive cohorts (of 3 patients) with different patients. Each cohort of patients will be closely monitored for one week before moving on to a new cohort. There will be no dose escalation in the same patient.
  The first 3 cohorts will use the mouthwash at 10%, 2, 3, and 4 times a day respectively. The last 3 cohorts will use the mouthwash at 15%, 2, 3, and 4 times a day respectively.
  If radiotherapy is interrupted for any reason and the patient is benefiting from using the mouthwash with copaiba, the patient will continue to perform the mouthwash.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Copaiba arm (Experimental): It will consist of the group of patients who will use copaiba mouthwash. It will be subdivided into 6 consecutive cohorts.
  Interventions: Drug: Copaiba

INTERVENTIONS:
Drug: Copaiba — A 10% and 15% aqueous solution of copaiba (Copaifera Officinalis Resin) manufactured by Interativo Farmácia de Manipulação will be used, under the formula: 10% copaiba oil (Copaifera Officinalis Resin) and 15% liquid mint aroma 5% , tween 80 1%, Aqueous solution (Distilled water + 0.1% Nipagin) qsp 100%.

SUMMARY:
This study aims to propose an alternative and auxiliary methodology for the prevention and treatment of Oral Mucositis (OM) in patients undergoing radiotherapy or radio and chemotherapy for head and neck neoplasms through the use of copaiba-based mouthwash, since the treatment that currently has proven efficacy for the prevention of OM(Low Power Laser Therapy) cannot be applied in tumor regions due to the risk of stimulating the tissue proliferation of malignant cells.

DETAILED DESCRIPTION:
This is a phase I study, carried out in a single institution to assess the safety and tolerability of using the aqueous copaiba solution for mouthwash in 03 to 36 patients diagnosed with cancer in the oral cavity.

In the selection/baseline period, the investigator or professional designated by him will assign a unique number to the patient being evaluated to participate in the study.

The investigator or professional designated by him may register the patient as soon as the eligibility for participation is confirmed and he signs the free and informed consent form. The patients included in the study will receive instructions on oral hygiene and the aqueous copaiba solution for mouthwash.

The recruitment and design of the study will be carried out according to the "3 + 3" design (modified Fibonacci design) with the planned inclusion of 6 successive cohorts (of 3 patients) with different patients. Each cohort of patients will be closely monitored for one week before moving on to a new cohort. There will be no dose escalation in the same patient. The concentration of the aqueous copaiba solution and the frequency of the mouthwash will be considered dose.

Patients will be treated according to the dose levels listed below, from the first day of radiation therapy:

* Cohort 1: 3 to 6 patients will be instructed to rinse with the solution 10% copaiba water, twice a day, for a period of 33 to 37 days*.
* Cohort 2: 3 to 6 patients will be instructed to rinse with the solution 10% copaiba water, 3 times a day, for a period of 33 to 37 days*.
* Cohort 3: 3 to 6 patients will be instructed to rinse with the solution 10% copaiba water, 4 times a day, for a period of 33 to 37 days*.
* Cohort 4: 3 to 6 patients will be instructed to rinse with the solution 15% copaiba water, twice a day, for a period of 33 to 37 days*.
* Cohort 5: 3 to 6 patients will be instructed to rinse with the solution 15% copaiba water, 3 times a day, for a period of 33 to 37 days*.
* Cohort 6: 3 to 6 patients will be instructed to rinse with the solution 15% copaiba water, 4 times a day, for a period of 33 to 37 days*.

  * If radiotherapy is interrupted for any reason and the patient is having benefit with the use of the copaiba mouthwash, the patient will continue the performance of the mouthwash during the period of interruption.
  * It will be admitted that in the D1 of radiotherapy/use of the copaiba mouthwash the patient performs only one of the mouthwashes described by the protocol.

Criteria for defining dose-limiting toxicity (DLT) Safety Safety assessments will be carried out by monitoring and recording all adverse events (AEs), including serious adverse events.

Adverse events For this protocol, an AE was defined as the appearance of undesirable medical signs, symptoms or conditions or worsening of existing ones, occurring from the signing of the informed consent form until the end of the study, even if the event is not considered as related to the interventions of the study.

AEs will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, except for the event of interest in this study - oral mucositis - which will be classified according to the Organization's oral mucositis scale World Health Organization (WHO).

The degree of OM according to the classification of the WHO of 1979, is subdivided into Degree 0 - No alteration (Absent); Grade 1 - Presence of erythema, Grade 2 - Presence of erythema and ulcers, but the patient can eat solid and liquid; Grade 3 - Presence of ulcers, but the patient can only eat a liquid and pasty diet and Grade 4 - Presence of ulcers and the ingestion of solids or liquids is impossible.

In this study, the criteria for defining DLT were established, as well as criteria for temporary interruptions of treatment with copaiba as described below.

Oral mucositis If oral mucositis grade 3 occurs in the first week of treatment in the tumor area, which will not be treated with laser therapy, treatment with copaiba will be interrupted for 1 week and symptomatic treatment with dipyrone and mouthwash with dexamethasone should be prescribed. If oral mucositis grade 4 occurs in the first week of treatment in the tumor area, which will not be treated with laser therapy, treatment with copaiba will be interrupted for 2 weeks and symptomatic treatment with dipyrone and mouthwash with dexamethasone should be prescribed. If the problem is resolved (or stabilized to a degree ≤ 2) within a maximum of 2 weeks, treatment may be restarted at the same dose level. If the problem persists for more than 2 consecutive weeks or 3 non-consecutive weeks, the respective patient should be discontinued from treatment (dose-limiting toxicity) and continue treatment with laser therapy, in areas not involved by the tumor, daily until the end of radiotherapy and with radiotherapy and cisplatin at the discretion of the attending physician.

If grade 2, 3, or 4 oral mucositis occurs after the second week of treatment in the tumor area, which will not be treated with laser therapy or in another region of the oral cavity receiving laser therapy, copaiba treatment will be maintained and treatment symptomatic with dipyrone or opioid should be prescribed.

Pain The pain will be classified according to CTCAE v5.0, associated with the Visual Analogue Scale, where a value of 0 corresponds to the absence of pain and 10, the greatest pain he can imagine. According to the standards established by the scale, values from 0 to 3 correspond to mild pain, from 4 to 6 to moderate pain, and from 7 to 10, severe pain.

In the absence of oral mucositis, if the patient reports pain in the grade 3 oral cavity, for the first time, in the first week of treatment in the tumor area, which will not be treated with laser therapy, the copaiba treatment will be interrupted for 1 week and one symptomatic dipyrone treatment should be prescribed. If pain in the grade 4 oral cavity occurs in the first week of treatment in the tumor area, which will not be treated with laser therapy, copaiba treatment will be interrupted for 2 weeks and symptomatic treatment with dipyrone or opioid should be prescribed.

In the absence of oral mucositis if the problem is resolved (or stabilized to a degree ≤ 2) within a maximum period of 2 weeks, treatment may be restarted at the same dose level. If the problem persists for more than 2 consecutive weeks or 3 non-consecutive weeks, the respective patient should be discontinued from treatment (toxicity limiting dose) and continue treatment with laser therapy, in areas not involved by the tumor, daily until the end of radiotherapy and with radiotherapy and cisplatin at the discretion of the attending physician.

In the presence of oral mucositis, the pain will not be considered dose-limiting toxicity (DLT), and if grade 2 or 3 oral pain occurs after the second week of treatment in the tumor area (which will not be treated with laser therapy) or in another region of the oral cavity receiving laser therapy, copaiba treatment will be maintained and symptomatic treatment with dipyrone or opioid should be prescribed.

If DLT is not observed in 3 patients at a given dose level, the dose will be escalated to the next level.

If the incidence of DLT is 33% (1 in 3 patients) 7 consecutive days, then 3 more patients will be treated with the same dose level. If DLT cases are not seen in these other 3 patients, then the dose will be escalated to the next level. Otherwise, the dose escalation will be stopped and recruitment will be terminated.

If the incidence of DLT is greater than 33% at a given level, then the dose escalation will be interrupted, the DLT will be defined as the maximum tolerated dose (MTD).

The patient will continue to be followed every two weeks (+/- 3 days) for eight weeks for safety assessment after the end of treatment with copaiba. Patients prematurely discontinued from the study treatment will only carry out the visit of discontinuation within seven days after the end of treatment. The end of treatment is defined such as the date of the safety assessment visit or discontinuation visit, whichever occurs first.

Radiotherapy and chemotherapy protocol

- Radiotherapy Radiotherapy (RT) will be performed according to the location of the tumor, using megavoltage radiotherapy with intensity-modulated radiotherapy techniques (IMRT). A total dose of 60 to 70 Gy will be applied daily between 30 to 35 fractions, 5 days a week, using IMRT or volumetrically modulated arc radiotherapy (VMAT).

The primary tumor and cervical lymph nodes will be treated with fields determined by imaging studies, with three-dimensional planning with image fusion (computed tomography, PET scan, or Resonance). The areas of macroscopic disease, as well as lymph node enlargement determined by images, will receive 70 Gy. The areas surrounding the injury will receive 59.4 Gy. The elective nodal areas will receive 56 Gy. In the case of postoperative adjuvant radiotherapy, the patient will receive 60 to 65 Gy according to the presence of compromised limits in the histopathological exam.

Radiation therapy will be suspended if patients present grade 4 dermatitis or weight loss greater than 10% and must be restarted after the clinical condition is restored, according to the protocol of the INCA Radiotherapy Service.

If the patient has a weight loss greater than 10%, he will receive nutritional support through a nasoenteral tube or gastrostomy.

- Chemotherapy Patients who have a clinical indication will be treated with cisplatin administered at a dose of 100mg / m², intravenously in 3 cycles of (more or less) 21 in 21 days.

Cisplatin will be suspended for one week if patients have grade 3 hematological toxicity, grade 2 nephrotoxicity, and grade 2 ototoxicity. In cases of grade 3 nephrotoxicity and grade 3 ototoxicity, cisplatin treatment will be discontinued, according to the protocol of the Clinical Oncology Section of INCA.

Oral hygiene protocol Patients will be instructed to perform oral hygiene after all meals, solid or liquid. In cases of exclusive use of a nasoenteral tube, patients will be instructed to brush their teeth three times a day. Oral hygiene will be performed with fluoridated toothpaste. From the tenth day of treatment with radiotherapy, patients will use an oral humidifying gel four times a day (Oral Balance®).

Low Power Laser Therapy The application of the LPLT will be carried out by the researcher responsible for the study in the Dentistry Section of INCA.

The assessment of the patient's oral mucosa will be performed by two dentists appointed by the principal investigator.

The application of the LPLT will start on the same day as the beginning of the RT and chemotherapy (CT), extending until the end of both and or the end of oral mucositis.

The application of LPLT will be performed daily, from Monday to Friday, before the radiotherapy session.

The application will be carried out with the DMC device (São Carlos, São Paulo, Brazil), with a gallium-aluminum indium phosphide diode (InGaAlP) with radiation emission in the red region of the electromagnetic spectrum (660 nm), with 100mW, with a beam area of 0.24cm². An energy of 1 J / point and an energy density of 4 J / cm² / point were determined, which will be applied punctually, with a distance between points of 1 cm, for 10s per point, totaling 9 points per region. A power meter (Handheld Laser Power Meeter (RoHS) will be used weekly to assess the condition of the device.

The treated regions of the oral mucosa will be: right and left cheek mucosa, lower and upper lip, upper and lower lip mucosa, right and left lateral border of the tongue, lingual belly, and buccal floor.

LPLT will not be performed in the tumor area. When patients have grade 2 oral mucositis, they will receive therapeutic LPLT with the energy of 2 J / point and energy density of 8 J / cm² / point.

Prevention of candidosis

Patients will use fluconazole 50 mg/day, orally, from Day 6 of radiotherapy until the end of it.

The aqueous solution of Copaiba

A 10% and 15% aqueous solution of copaiba (Copaifera Officinalis Resin) manufactured by Interativo Farmácia de Manipulação will be used, under the formula: 10% copaiba oil (Copaifera Officinalis Resin) and 15% liquid mint aroma 5% , tween 80 1%, Aqueous solution (Distilled water + 0.1% Nipagin) qsp 100%.

The product will be stored at room temperature and will be stored in the Dentistry Section of INCA.

Data collect

Patient data will be collected from physical and electronic medical records and will be transcribed to the specific clinical record of the study. The data of interest are age, sex (female and male), the education level (illiterate, elementary, middle and higher, complete or incomplete), underlying disease, the treatment used for the disease, with specification on the type of chemotherapy and radiotherapy performed, the dose received and fractionation, presence of associated comorbidities, adverse events, and data related to physical examination during the study. The presence of habits such as smoking and alcohol consumption (duration of the habit, daily amount, if the habit was abandoned or not; if so, for how long) will also be recorded. The data will be included in REDCap®, an electronic data collection system, in forms customized for this research project.

- Dental Evaluation

Patients will undergo daily intraoral physical examination from the beginning to the end of treatment, using the research form. Sialometry will be assessed weekly.

The mucous membranes will be evaluated for their color, hydration, integrity, presence of OM. The characteristics of pseudomembranous and erythematous candidiasis according to Neville will be considered signs of fungal infection. Pseudomembranous candidiasis appears in the form of white, creamy, detachable plaques and halitosis, while the erythematosus appears as red spots. Viral infections will be classified as those that present as multiple small and erythematous papules, which form clusters of liquid-filled vesicles, which break, forming ulcers in the sequence forming crusts within 2 days, thus characterizing herpes simplex.

The degree of OM will be established according to the classification of the World Health Organization (WHO) of 1979, which subdivides it into Degree 0 - No alteration (Absent); Grade 1 - Presence of erythema, Grade 2 - Presence of erythema and ulcers, but the patient can eat solid and liquid; Grade 3 - Presence of ulcers, but the patient can only eat a liquid and pasty diet and Grade 4 - Presence of ulcers and the ingestion of solids or liquids is impossible.

The investigators will also use the criteria established by Sonis et al in 1999, which considers the presence and size of ulcerations/pseudomembranes and erythema. Ulcerations/pseudomembranes will be assessed in the following scores: 0 - in the absence of lesions, 1 - in lesions smaller than 1 cm3, 2 - in lesions measuring between 1 and 3 cm3, and 3 - in lesions larger than 3 cm3. Erythema will be evaluated according to the following scores: 0 - when absent, 1 - when present, but not severe, and 2 - when present and severe.

On the Sonis scale, the daily calculation of the sum of the weighted average of the ulcerated area and the intensity of the erythema (MP = 2.5 x [(∑ui: 3 x Nu) + (∑ei: 2 x Ne)] will be performed, where ∑ ui = sum of the ulcerated area, Nu = number of ulcerated areas, ∑ei = sum of the erythema intensity and Ne = number of areas with erythema. A millimeter dental ruler was used to measure the area.

Since xerostomia is the term used to describe a subjective condition of dry mouth sensation due to the absence of saliva, the assessment of this item will be made according to the presence of the complaint about this condition or not by the patient, associated sialometry according to CTCAE v5.0.

Regarding pain, patients will be asked about its presence or absence. The pain will be classified according to CTCAE v5.0, associated with the Visual Analogue Scale, where a value of 0 corresponds to the absence of pain and 10, the greatest pain he can imagine. According to the standards established by the scale, values from 0 to 3 correspond to mild pain, from 4 to 6 to moderate pain, and from 7 to 10, severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients enrolled at INCA with a diagnosis of cell carcinoma squamous, adenoid cystic carcinoma, mucoepidermoid carcinoma, carcinoma of acinar cells, low-grade polymorph adenocarcinoma, located in the oral cavity (ICD-10 C00 to C06); located in the oral cavity with the indication of exclusive radiotherapy (by IMRT/VMAT technique) or radiotherapy (by IMRT/ VMAT) associated with chemotherapy.
* Performance status (PS) 0 or 1.
* Patients with intact oral mucosa (except the tumor area) without color change and volume on the first day of treatment.
* Patients able to cooperate with treatment.
* Patients capable of performing the oral hygiene protocol.
* Patients who after the information and instructions signed the term of free and informed consent of the patient in accordance with Resolution 466/12 of the National Health Council.

Exclusion Criteria:

* Patients who are receiving drugs for the treatment and/or prevention of oral mucositis.
* Patients undergoing radiotherapy with planning that excludes the oral cavity of the treatment field.
* Patients undergoing palliative radiotherapy.
* Patients with cervical lymph node metastasis greater than 6cm (N3).
* Patients who report any type of allergy to copaiba-based compounds.
* Patients diagnosed with oral lichen planus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2025-09-07 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Through the use of the copaiba oil, an average of 6 to 7 weeks.
  Evaluate the maximum tolerated dose of the aqueous copaiba solution.

SECONDARY OUTCOMES:
Acess rate of pain | From baseline to the last day of copaiba use (day 33 to day 37).
  Assess the level of pain of the patients during the mouthwash with the aqueous copaiba solution through the visual analog pain scale (classified between 0 to 10, when a higher score means worst level of pain)
Acess rate of oral pain | From baseline to the last day of copaiba use (day 33 to day 37).
  Assess the level of pain of the patients during the mouthwash with the aqueous copaiba solution through the criteria proposed by the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0.(classified between grades 1 to 3, when a higher score means worst level of pain)
Incidence of Oral Mucositis | From baseline to the last day of copaiba use (day 33 to day 37).
  Check the incidence of oral mucositis in the treated and untreated areas with low power laser.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
Data will be released after the study is completed.

REFERENCES:
- [Background] Addy M. Oral hygiene products: potential for harm to oral and systemic health? Periodontol 2000. 2008;48:54-65. doi: 10.1111/j.1600-0757.2008.00253.x. No abstract available. PMID 18715356
- [Background] Ames-Sibin AP, Barizao CL, Castro-Ghizoni CV, Silva FMS, Sa-Nakanishi AB, Bracht L, Bersani-Amado CA, Marcal-Natali MR, Bracht A, Comar JF. beta-Caryophyllene, the major constituent of copaiba oil, reduces systemic inflammation and oxidative stress in arthritic rats. J Cell Biochem. 2018 Dec;119(12):10262-10277. doi: 10.1002/jcb.27369. Epub 2018 Aug 21. PMID 30132972
- [Background] Antunes HS, Herchenhorn D, Small IA, Araujo CM, Viegas CM, Cabral E, Rampini MP, Rodrigues PC, Silva TG, Ferreira EM, Dias FL, Ferreira CG. Phase III trial of low-level laser therapy to prevent oral mucositis in head and neck cancer patients treated with concurrent chemoradiation. Radiother Oncol. 2013 Nov;109(2):297-302. doi: 10.1016/j.radonc.2013.08.010. Epub 2013 Sep 14. PMID 24044799
- [Background] Antunes HS, de Azevedo AM, da Silva Bouzas LF, Adao CA, Pinheiro CT, Mayhe R, Pinheiro LH, Azevedo R, D'Aiuto de Matos V, Rodrigues PC, Small IA, Zangaro RA, Ferreira CG. Low-power laser in the prevention of induced oral mucositis in bone marrow transplantation patients: a randomized trial. Blood. 2007 Mar 1;109(5):2250-5. doi: 10.1182/blood-2006-07-035022. Epub 2006 Oct 19. PMID 17053058
- [Background] Antunes HS, Ferreira EM, de Faria LM, Schirmer M, Rodrigues PC, Small IA, Colares M, Bouzas LF, Ferreira CG. Streptococcal bacteraemia in patients submitted to hematopoietic stem cell transplantation: the role of tooth brushing and use of chlorhexidine. Med Oral Patol Oral Cir Bucal. 2010 Mar 1;15(2):e303-9. doi: 10.4317/medoral.15.e303. PMID 20038916
- [Background] Ariyawardana A, Cheng KKF, Kandwal A, Tilly V, Al-Azri AR, Galiti D, Chiang K, Vaddi A, Ranna V, Nicolatou-Galitis O, Lalla RV, Bossi P, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society for Oral Oncology (MASCC/ISOO). Systematic review of anti-inflammatory agents for the management of oral mucositis in cancer patients and clinical practice guidelines. Support Care Cancer. 2019 Oct;27(10):3985-3995. doi: 10.1007/s00520-019-04888-w. Epub 2019 Jul 8. PMID 31286230
- [Background] Bensadoun RJ, Franquin JC, Ciais G, Darcourt V, Schubert MM, Viot M, Dejou J, Tardieu C, Benezery K, Nguyen TD, Laudoyer Y, Dassonville O, Poissonnet G, Vallicioni J, Thyss A, Hamdi M, Chauvel P, Demard F. Low-energy He/Ne laser in the prevention of radiation-induced mucositis. A multicenter phase III randomized study in patients with head and neck cancer. Support Care Cancer. 1999 Jul;7(4):244-52. doi: 10.1007/s005200050256. PMID 10423050
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Cohen N, Fedewa S, Chen AY. Epidemiology and Demographics of the Head and Neck Cancer Population. Oral Maxillofac Surg Clin North Am. 2018 Nov;30(4):381-395. doi: 10.1016/j.coms.2018.06.001. Epub 2018 Aug 3. PMID 30078696
- [Background] Dalenogare DP, Ferro PR, De Pra SDT, Rigo FK, de David Antoniazzi CT, de Almeida AS, Damiani AP, Strapazzon G, de Oliveira Sardinha TT, Galvani NC, Boligon AA, de Andrade VM, da Silva Brum E, Oliveira SM, Trevisan G. Antinociceptive activity of Copaifera officinalis Jacq. L oil and kaurenoic acid in mice. Inflammopharmacology. 2019 Aug;27(4):829-844. doi: 10.1007/s10787-019-00588-3. Epub 2019 May 16. PMID 31098702
- [Background] Dias-da-Silva MA, Pereira AC, Marin MC, Salgado MA. The influence of topic and systemic administration of copaiba oil on the alveolar wound healing after tooth extraction in rats. J Clin Exp Dent. 2013 Oct 1;5(4):e169-73. doi: 10.4317/jced.51104. eCollection 2013 Oct 1. PMID 24455075
- [Background] Diefenbach AL, Muniz FWMG, Oballe HJR, Rosing CK. Antimicrobial activity of copaiba oil (Copaifera ssp.) on oral pathogens: Systematic review. Phytother Res. 2018 Apr;32(4):586-596. doi: 10.1002/ptr.5992. Epub 2017 Nov 29. PMID 29193389
- [Background] Estevao LR, Medeiros JP, Baratella-Evencio L, Simoes RS, Mendonca Fde S, Evencio-Neto J. Effects of the topical administration of copaiba oil ointment (Copaifera langsdorffii) in skin flaps viability of rats. Acta Cir Bras. 2013 Dec;28(12):863-9. doi: 10.1590/s0102-86502013001200009. PMID 24316860
- [Background] Fidler P, Loprinzi CL, O'Fallon JR, Leitch JM, Lee JK, Hayes DL, Novotny P, Clemens-Schutjer D, Bartel J, Michalak JC. Prospective evaluation of a chamomile mouthwash for prevention of 5-FU-induced oral mucositis. Cancer. 1996 Feb 1;77(3):522-5. doi: 10.1002/(SICI)1097-0142(19960201)77:33.0.CO;2-6. PMID 8630960
- [Background] Gelmini F, Beretta G, Anselmi C, Centini M, Magni P, Ruscica M, Cavalchini A, Maffei Facino R. GC-MS profiling of the phytochemical constituents of the oleoresin from Copaifera langsdorffii Desf. and a preliminary in vivo evaluation of its antipsoriatic effect. Int J Pharm. 2013 Jan 20;440(2):170-8. doi: 10.1016/j.ijpharm.2012.08.021. Epub 2012 Aug 20. PMID 22939967
- [Background] Gomes Nde M, de Rezende CM, Fontes SP, Matheus ME, Pinto Ada C, Fernandes PD. Characterization of the antinociceptive and anti-inflammatory activities of fractions obtained from Copaifera multijuga Hayne. J Ethnopharmacol. 2010 Mar 2;128(1):177-83. doi: 10.1016/j.jep.2010.01.005. Epub 2010 Jan 12. PMID 20064592
- [Background] Gooi Z, Fakhry C, Goldenberg D, Richmon J, Kiess AP; Education Committee of the American Head and Neck Society (AHNS). AHNS Series: Do you know your guidelines?Principles of radiation therapy for head and neck cancer: A review of the National Comprehensive Cancer Network guidelines. Head Neck. 2016 Jul;38(7):987-92. doi: 10.1002/hed.24448. Epub 2016 Mar 25. PMID 27015108
- [Background] GUTKNECHT, N.; EDUARDO, C. P. A odontologia e o laser. Primeira e ed. [s.l.]: Berlin: Quintessence, 2004. 25-60 p.
- [Background] INCA. Estimativa 2020: incidêcia de câncer no Brasil. [s.l.]: Instituto Nacional de Câncer José Alencar Gomes da Silva/ Ministério da Saúde, 2019. ISBN: 9788573183887.
- [Background] Jones JA, Avritscher EB, Cooksley CD, Michelet M, Bekele BN, Elting LS. Epidemiology of treatment-associated mucosal injury after treatment with newer regimens for lymphoma, breast, lung, or colorectal cancer. Support Care Cancer. 2006 Jun;14(6):505-15. doi: 10.1007/s00520-006-0055-4. Epub 2006 Apr 7. PMID 16601950
- [Background] Lalla RV, Bowen J, Barasch A, Elting L, Epstein J, Keefe DM, McGuire DB, Migliorati C, Nicolatou-Galitis O, Peterson DE, Raber-Durlacher JE, Sonis ST, Elad S; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2014 May 15;120(10):1453-61. doi: 10.1002/cncr.28592. Epub 2014 Feb 25. PMID 24615748
- [Background] Leandro LM, Vargas Fde S, Barbosa PC, Neves JK, da Silva JA, da Veiga-Junior VF. Chemistry and biological activities of terpenoids from copaiba (Copaifera spp.) oleoresins. Molecules. 2012 Mar 30;17(4):3866-89. doi: 10.3390/molecules17043866. PMID 22466849
- [Background] Lima CS, de Medeiros BJ, Favacho HA, dos Santos KC, de Oliveira BR, Taglialegna JC, da Costa EV, de Campos KJ, Carvalho JC. Pre-clinical validation of a vaginal cream containing copaiba oil (reproductive toxicology study). Phytomedicine. 2011 Sep 15;18(12):1013-23. doi: 10.1016/j.phymed.2011.05.004. Epub 2011 Jun 12. PMID 21665449
- [Background] Lydiatt WM, Patel SG, O'Sullivan B, Brandwein MS, Ridge JA, Migliacci JC, Loomis AM, Shah JP. Head and Neck cancers-major changes in the American Joint Committee on cancer eighth edition cancer staging manual. CA Cancer J Clin. 2017 Mar;67(2):122-137. doi: 10.3322/caac.21389. Epub 2017 Jan 27. PMID 28128848
- [Background] Marur S, Forastiere AA. Head and Neck Squamous Cell Carcinoma: Update on Epidemiology, Diagnosis, and Treatment. Mayo Clin Proc. 2016 Mar;91(3):386-96. doi: 10.1016/j.mayocp.2015.12.017. PMID 26944243
- [Background] Mazokopakis EE, Vrentzos GE, Papadakis JA, Babalis DE, Ganotakis ES. Wild chamomile (Matricaria recutita L.) mouthwashes in methotrexate-induced oral mucositis. Phytomedicine. 2005 Jan;12(1-2):25-7. doi: 10.1016/j.phymed.2003.11.003. PMID 15693704
- [Background] MENEZES, A. C. et al. Abordagem clínica e terapêutica da mucosite oral induzida por radioterapia e quimioterapia em pacientes com câncer. Revistas, [s.l.], v. 71, no 1, p. 35, 2014. ISSN: 0034-7272, DOI: 10.18363/rbo.v71i1.536.
- [Background] Mifsud M, Eskander A, Irish J, Gullane P, Gilbert R, Brown D, de Almeida JR, Urbach DR, Goldstein DP. Evolving trends in head and neck cancer epidemiology: Ontario, Canada 1993-2010. Head Neck. 2017 Sep;39(9):1770-1778. doi: 10.1002/hed.24829. Epub 2017 May 30. PMID 28557276
- [Background] Migliorati C, Hewson I, Lalla RV, Antunes HS, Estilo CL, Hodgson B, Lopes NN, Schubert MM, Bowen J, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of laser and other light therapy for the management of oral mucositis in cancer patients. Support Care Cancer. 2013 Jan;21(1):333-41. doi: 10.1007/s00520-012-1605-6. Epub 2012 Sep 22. PMID 23001179
- [Background] NEVILLE, B. W. et al. Patologia Oral e Maxilofacial. Terceira E ed. Rio de Janeiro: Elsevier, 2012. ISBN: 9788535230895.
- [Background] Pfeifer Barbosa AL, Wenzel-Storjohann A, Barbosa JD, Zidorn C, Peifer C, Tasdemir D, Cicek SS. Antimicrobial and cytotoxic effects of the Copaifera reticulata oleoresin and its main diterpene acids. J Ethnopharmacol. 2019 Apr 6;233:94-100. doi: 10.1016/j.jep.2018.11.029. Epub 2018 Nov 23. PMID 30472403
- [Background] PIERI, F. A.; MUSSI, M. C.; MOREIRA, M. A. S. Óleo de copaíba (Copaifera sp.): Histórico, extração, aplicações industrials e propriedades medicinais. Revista Brasileira de Plantas Medicinais, [s.l.], v. 11, no 4, p. 465-472, 2009. ISSN: 15160572, DOI: 10.1590/s1516-05722009000400016.
- [Background] Pieri FA, Mussi MC, Fiorini JE, Moreira MA, Schneedorf JM. Bacteriostatic effect of copaiba oil (Copaifera officinalis) against Streptococcus mutans. Braz Dent J. 2012;23(1):36-8. doi: 10.1590/s0103-64402012000100006. PMID 22460312
- [Background] Pinna R, Campus G, Cumbo E, Mura I, Milia E. Xerostomia induced by radiotherapy: an overview of the physiopathology, clinical evidence, and management of the oral damage. Ther Clin Risk Manag. 2015 Feb 4;11:171-88. doi: 10.2147/TCRM.S70652. eCollection 2015. PMID 25691810
- [Background] Rettig EM, D'Souza G. Epidemiology of head and neck cancer. Surg Oncol Clin N Am. 2015 Jul;24(3):379-96. doi: 10.1016/j.soc.2015.03.001. Epub 2015 Apr 9. PMID 25979389
- [Background] Ricardo LM, Dias BM, Mugge FLB, Leite VV, Brandao MGL. Evidence of traditionality of Brazilian medicinal plants: The case studies of Stryphnodendron adstringens (Mart.) Coville (barbatimao) barks and Copaifera spp. (copaiba) oleoresin in wound healing. J Ethnopharmacol. 2018 Jun 12;219:319-336. doi: 10.1016/j.jep.2018.02.042. Epub 2018 Mar 2. PMID 29501844
- [Background] Sahebjamee M, Mansourian A, Hajimirzamohammad M, Zadeh MT, Bekhradi R, Kazemian A, Manifar S, Ashnagar S, Doroudgar K. Comparative Efficacy of Aloe vera and Benzydamine Mouthwashes on Radiation-induced Oral Mucositis: A Triple-blind, Randomised, Controlled Clinical Trial. Oral Health Prev Dent. 2015;13(4):309-15. doi: 10.3290/j.ohpd.a33091. PMID 25431805
- [Background] SCHIRMER, E. M.; FERRARI, A.; TRINDADE, L. C. T. Evolução da mucosite oral após intervenção nutricional em pacientes oncológicos no serviço de cuidados paliativos. Revista Dor, [s.l.], v. 13, no 2, p. 141-146, 2012. ISSN: 2317-6393, DOI: 10.1590/s1806-00132012000200009.
- [Background] Scully C, Epstein J, Sonis S. Oral mucositis: a challenging complication of radiotherapy, chemotherapy, and radiochemotherapy. Part 2: diagnosis and management of mucositis. Head Neck. 2004 Jan;26(1):77-84. doi: 10.1002/hed.10326. PMID 14724910
- [Background] Simoes CA, Conde NC, Venancio GN, Milerio PS, Bandeira MF, da Veiga Junior VF. Antibacterial Activity of Copaiba Oil Gel on Dental Biofilm. Open Dent J. 2016 May 11;10:188-95. doi: 10.2174/1874210601610010188. eCollection 2016. PMID 27386004
- [Background] Sonis ST, Eilers JP, Epstein JB, LeVeque FG, Liggett WH Jr, Mulagha MT, Peterson DE, Rose AH, Schubert MM, Spijkervet FK, Wittes JP. Validation of a new scoring system for the assessment of clinical trial research of oral mucositis induced by radiation or chemotherapy. Mucositis Study Group. Cancer. 1999 May 15;85(10):2103-13. doi: 10.1002/(sici)1097-0142(19990515)85:103.0.co;2-0. PMID 10326686
- [Background] Sonis ST, Elting LS, Keefe D, Peterson DE, Schubert M, Hauer-Jensen M, Bekele BN, Raber-Durlacher J, Donnelly JP, Rubenstein EB; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Perspectives on cancer therapy-induced mucosal injury: pathogenesis, measurement, epidemiology, and consequences for patients. Cancer. 2004 May 1;100(9 Suppl):1995-2025. doi: 10.1002/cncr.20162. PMID 15108222
- [Background] Sonis ST. Mucositis: The impact, biology and therapeutic opportunities of oral mucositis. Oral Oncol. 2009 Dec;45(12):1015-20. doi: 10.1016/j.oraloncology.2009.08.006. Epub 2009 Oct 13. PMID 19828360
- [Background] Sroussi HY, Jessri M, Epstein J. Oral Assessment and Management of the Patient with Head and Neck Cancer. Oral Maxillofac Surg Clin North Am. 2018 Nov;30(4):445-458. doi: 10.1016/j.coms.2018.06.006. Epub 2018 Aug 31. PMID 30173900
- [Background] Tobouti PL, de Andrade Martins TC, Pereira TJ, Mussi MCM. Antimicrobial activity of copaiba oil: A review and a call for further research. Biomed Pharmacother. 2017 Oct;94:93-99. doi: 10.1016/j.biopha.2017.07.092. Epub 2017 Jul 27. PMID 28756369
- [Background] da Trindade R, da Silva JK, Setzer WN. Copaifera of the Neotropics: A Review of the Phytochemistry and Pharmacology. Int J Mol Sci. 2018 May 18;19(5):1511. doi: 10.3390/ijms19051511. PMID 29783680
- [Background] Valadas LAR, Gurgel MF, Mororo JM, Fonseca SGDC, Fonteles CSR, de Carvalho CBM, Fechine FV, Rodrigues Neto EM, de Franca Fonteles MM, Chagas FO, Lobo PLD, Bandeira MAM. Dose-response evaluation of a copaiba-containing varnish against streptococcus mutans in vivo. Saudi Pharm J. 2019 Mar;27(3):363-367. doi: 10.1016/j.jsps.2018.12.004. Epub 2018 Dec 15. PMID 30976179
- [Background] Wagner VP, Webber LP, Ortiz L, Rados PV, Meurer L, Lameira OA, Lima RR, Martins MD. Effects of Copaiba Oil Topical Administration on Oral Wound Healing. Phytother Res. 2017 Aug;31(8):1283-1288. doi: 10.1002/ptr.5845. Epub 2017 Jun 21. PMID 28635033
- [Background] Yarom N, Ariyawardana A, Hovan A, Barasch A, Jarvis V, Jensen SB, Zadik Y, Elad S, Bowen J, Lalla RV; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of natural agents for the management of oral mucositis in cancer patients. Support Care Cancer. 2013 Nov;21(11):3209-21. doi: 10.1007/s00520-013-1869-5. Epub 2013 Jun 14. PMID 23764678
- [Background] Zadik Y, Arany PR, Fregnani ER, Bossi P, Antunes HS, Bensadoun RJ, Gueiros LA, Majorana A, Nair RG, Ranna V, Tissing WJE, Vaddi A, Lubart R, Migliorati CA, Lalla RV, Cheng KKF, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of photobiomodulation for the management of oral mucositis in cancer patients and clinical practice guidelines. Support Care Cancer. 2019 Oct;27(10):3969-3983. doi: 10.1007/s00520-019-04890-2. Epub 2019 Jul 8. PMID 31286228
- [Background] INCA, I. N. de C. Cuidados paliativos oncológicos. Cuidados Paliativos Oncológicos. [s.l.]: [s.n.], 2001. v. 22, 2055-2066 p. ISBN: 857318079X